CLINICAL TRIAL: NCT03756662
Title: A Prospective, Open-label, Single Arm, Multicenter Clinical Investigation to Assess the Safety and Performance of the ARGOS-SC Suprachoroidal Pressure Sensor System in Patients With Glaucoma Undergoing Non-penetrating Glaucoma Surgery
Brief Title: Performance and Safety of the ARGOS-SC Suprachoroidal Pressure Sensor in Patients With Glaucoma Undergoing Non-penetrating Glaucoma Surgery
Acronym: ARGOS-SC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implandata Ophthalmic Products GmbH (Industry)
Collaborators: CRO Dr. med Kottmann GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARGOS-SC01; CIV-18-07-025065 (Registry Identifier: Eudamed)
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma; Open Angle Glaucoma
Keywords: Non-penetrating glaucoma surgery; Open angle glaucoma; Intraocular pressure measurements; Suprachoroidal pressure sensor; ARGOS-SC
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single arm, multicenter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARGOS-SC Sensor (Experimental): In this prospective, multicenter, open-label, single-arm, interventional clinical trial, 24 eyes of 24 POAG patients who were due to undergo NPGS (canaloplasty or deep sclerectomy) were enrolled. An ARGOS-SC sensor was implanted during NPGS. Goldmann applanation tonometry (GAT) measures were compared with the sensors' IOP measures at all post-operative visits through 12 months. Device position and adverse events were recorded throughout the follow-up.
  Interventions: Device: ARGOS-SC suprachoroidal pressure sensor

INTERVENTIONS:
Device: ARGOS-SC suprachoroidal pressure sensor — The sensor device is intended to be permanently implanted suprachoroidal in the human eye during non-penetrating glaucoma surgery.

SUMMARY:
The purpose of this study is to evaluate both the safety and feasibility of the surgical implantation of the ARGOS-SC implant during non-penetrating glaucoma surgery and the safety and usability of the ARGOS-SC implant and system in the year following the implantation.

DETAILED DESCRIPTION:
This study is designed as a prospective, open-label, multicenter, single-arm clinical investigation. Subjects will be followed up at regular intervals for one year following implantation to collect safety and performance information. Enrollment will be halted at every serious adverse device event (SADE).

The sensor device is intended to be permanently implanted suprachoroidal in the human eye during non-penetrating glaucoma surgery and is used in conjunction with the hand-held MESOGRAPH reading device to telemetrically measure the intraocular pressure (IOP) of the implanted eye.

The sample size calculation was based on the study's dual purpose of establishing safety and comparability of IOP measurements with the ARGOS-SC system to those made with GAT and DCT. IOP measurements will be made with all devices at various time points, resulting in a within individual control for IOP variables. Based on these calculations (performance, safety) and considering possible drop-outs, the exploratory investigation will enroll 24 patients. The minimum number of measurements required to hold the performance claim is approx. 120. With multiple (>8) measurements with either method (ARGOS, GAT) per patient, a sufficient number of paired measurements (in total >>120 measurement pairs) will be available to show equivalence of the methods (primary objective).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to understand the informed consent and willing to participate as evidenced by providing informed consent.
2. Male or female aged ≥ 18 years on the day of screening Female subjects of childbearing potential (not surgically sterilized or more than one year post-menopausal) must be willing to use adequate contraception throughout the trial and must have a negative pregnancy test (urine beta-hCG) within 24 hours prior to ARGOS-SC pressure sensor implantation.
3. Diagnosis of open angle glaucoma requiring a non-penetrating glaucoma surgery (NPGS). The medical indication for a non-penetrating glaucoma surgery must be given irrespective of the study participation. Potential study patients will be solicited for participation in the clinical trial only after the patient has given consent to the non-penetrating glaucoma operation.
4. Subjects able and willing to attend all scheduled visits and comply with all study procedures

Exclusion Criteria:

1. Contraindications for a non-penetrating glaucoma surgery

   * Neovascular glaucoma, primary and secondary angle closure glaucoma
   * Condition after previous glaucoma incisional surgery
   * IOP > 40 mmHg
2. Myopia (> -6 dpt) or hypermetropia (> +4 dpt)
3. Axis length < 22 mm or > 26 mm
4. Exudative age-related macular degeneration, instable macular degeneration 30 days prior to inclusion, or macular edema
5. Acute retinal detachment
6. Uncontrolled Diabetes Mellitus (DM) with manifestation of moderate to severe non-proliferative diabetic Retinopathy (DR) or proliferative DR.
7. History or evidence of severe active inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to ARGOS-SC implantation
8. Ocular surgery procedure(s) (excluding selective laser trabeculoplasty and peripheral iridotomy) within 6 months (cataract surgery within 3 months) prior to ARGOS-SC implantation in the study eye that can affect the assessment of IOP by Goldmann Applanation tonometry
9. Ocular disease other than glaucoma that may affect assessment of visual acuity and/or IOP by Goldmann Applanation tonometry/Pascal Dynamic Contour Tonometry (e.g. choroidal hemorrhage or detachment, lens subluxation, thyroid ophthalmopathy)
10. Existence of other active medical eye implant and/or other active medical implants in the head/neck region
11. Difficulties or complications during NPGS procedure or implantation of ARGOS-SC sensor, as assessed by surgeon (e.g. perforation of trabeculo-descement's membrane; excessive aqueous filtration through TDM leading to shallow anterior chamber; excessive bleeding; choroidal detachment)
12. Severe generalized disease resulting in a life expectancy shorter than a year
13. Currently pregnant or breastfeeding
14. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device
15. Patients who are not suitable for the study based on the surgeon's evaluation
16. Patients unable or unwilling to understand or comply with required study procedures
17. Patients with psychiatric disorders influencing their judgement or autonomy
18. Subject and/or an immediate family member is an employee of the investigational site directly affiliated with this study, the sponsor or the contract research organization.
19. Enrollment of the fellow eye in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szurman, Prof., Principal Investigator — Knappschaftsklinikum Saar GmbH, Augenklinik Sulzbach
Locations (5):
- Germany (4):
  - Universitäts-Augenklinik, Bochum
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Augenklinik und Poliklinik, Mainz
  - Augenklinik der LMU München, München
  - Knappschaftsklinikum Saar GmbH, Augenklinik Sulzbach, Sulzbach
- Swiss Glaucoma Research Foundation, Centre du Glaucome, Clinique Montchoisi, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szurman P, Gillmann K, Seuthe AM, Dick HB, Hoffmann EM, Mermoud A, Mackert MJ, Weinreb RN, Rao HL, Mansouri K; EYEMATE-SC Study Group. EYEMATE-SC Trial: Twelve-Month Safety, Performance, and Accuracy of a Suprachoroidal Sensor for Telemetric Measurement of Intraocular Pressure. Ophthalmology. 2023 Mar;130(3):304-312. doi: 10.1016/j.ophtha.2022.09.021. Epub 2022 Oct 3. PMID 36202141
- [Derived] Szurman P, Mansouri K, Dick HB, Mermoud A, Hoffmann EM, Mackert M, Weinreb RN, Rao HL, Seuthe AM; EYEMATE-SC study group. Safety and performance of a suprachoroidal sensor for telemetric measurement of intraocular pressure in the EYEMATE-SC trial. Br J Ophthalmol. 2023 Apr;107(4):518-524. doi: 10.1136/bjophthalmol-2021-320023. Epub 2021 Nov 12. PMID 34772665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from November 2018 to January 2020 in medical clinics.
Groups:
- ARGOS-SC Sensor: In this prospective, multicenter, open-label, single-arm, interventional clinical trial, 24 eyes of 24 POAG patients who were due to undergo NPGS (canaloplasty or deep sclerectomy) were enrolled. An ARGOS-SC sensor was implanted during NPGS. Goldmann applanation tonometry(GAT) measures were compared with the sensors' IOP measures and comprehensive ophthalmic examinations at all post-operative visits (V02-V09) through 12 months. Device position and adverse events were recorded throughout the follow-up.
Period: Overall Study
Arm/Group | ARGOS-SC Sensor
Started | 24
Completed | 23
Not Completed | 1
Not completed — due to an SAE that was not related to the medical device or medical procedure. | 1

BASELINE CHARACTERISTICS:
Groups:
- ARGOS-SC Sensor: In this prospective, multicenter, open-label, single-arm, interventional clinical trial, 24 eyes of 24 POAG patients who were due to undergo NPGS (canaloplasty or deep sclerectomy) were enrolled. An ARGOS-SC sensor was implanted during NPGS. Goldmann applanation tonometry (GAT) measures were compared with the sensors' IOP measures and comprehensive ophthalmic examinations at all post-operative visits (V02-V09) through 12 months. Device position and adverse events were recorded throughout the follow-up.
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 4
  Germany | 20
Type of Glaucoma [Count of Participants; unit: Participants]
  Primary open-angle glaucoma (POAG) | 17
  Ocular hypertension (OHT)/Glaucoma suspect | 2
  Pseudoexfoliative (PEX) glauoma | 2
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Performance: Level of Agreement Between GAT and the ARGOS-SC System
Description: Level of Agreement between intraocular pressure (IOP) measurements made using GAT & the ARGOS-SC system (IOP in mmHg) following the Bland-Altman method.
Time Frame: Day 1 to Day 360 (V02 to V09)
Population: All available GAT and ARGOS-SC measurements.
Measure: Mean (95% Confidence Interval); unit: mmHg
Units Other Than Participants: comparisons
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 24
Number analyzed (comparisons) | 536
mmHg
  Overall Level of Agreement | 0.8 [-5.1 to 6.7]
  Level of Agreement 3-month post-operatively until the end of the follow-up | -0.2 [-4.6 to 4.2]

2. Secondary Outcome: Safety: Number of Patients Experiencing a Device-related SAE (SADE)
Description: Number of patients experiencing a device-related SAE (SADE).
Time Frame: Day 0 to Day 360 (V01 [Implantation] to V09)
Measure: Number; unit: participants
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 24
participants | 0

3. Secondary Outcome: Safety: Incidence, Nature, Severity and Seriousness of Observed Adverse Events (AEs) and Adverse Device Events (ADEs)
Description: Safety evaluation based on the incidence, nature, severity and seriousness of observed adverse events and adverse device events.
Time Frame: Day 0 to Day 360 (V01 [Implantation] to V09)
Population: A total of 98 AEs in 22 patients were reported in the ARGOS-SC study. In overall 54 adverse events were documented in 20 patients affecting the study eye. 11 out of 98 AEs in 7 Patients fulfilled at least one criterion for "serious adverse event" (SAE) and were reported as such. All of these SAEs were unrelated to the medical device or implantation procedure.
Measure: Number; unit: A(D)Es
Units Other Than Participants: Total number of AEs
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 24
Number analyzed (Total number of AEs) | 98
A(D)Es
  Overall number of AEs/ADEs affecting the study eye, of which | 54
  AEs related to medical procedure and/or | 44
  AEs related to medical device and/or | 16
  AEs related to other | 7

4. Secondary Outcome: Performance: Percentage of Measurements Within +/- 5 mmHg
Description: Concordance of the ARGOS-SC<>GAT measurement. Method applied: The probability distribution of the difference in the measurements made using GAT & the ARGOS-SC system per visit ("paired measurement") grouped within 1 mmHg was compared to the outcome measure of achieving 70% agreement of the total number of comparisons between +/-5 mmHg. The first column presents the overall data and the second column presents data from 3 months postoperatively onwards.
Time Frame: Day 1 to Day 360 (V02 to V09)
Population: All available GAT<>ARGOS-SC comparisons.
Measure: Number; unit: percentage of measurements
Units Other Than Participants: comparisons
Groups:
- ARGOS-SC Sensor: Comparisons between ARGOS-SC and GAT at all post-operative visits (V02-V09) through 12 months.
- ARGOS-SC Sensor After 3 Month Postoperative: Comparisons between ARGOS-SC and GAT at post-operative visits (V05-V09) 3 month through 12 month.
Arm/Group | ARGOS-SC Sensor | ARGOS-SC Sensor After 3 Month Postoperative
Number analyzed (Participants) | 24 | 24
Number analyzed (comparisons) | 181 | 87
percentage of measurements | 91 | 98

5. Secondary Outcome: Performance: Device Malfunctions
Description: Incidence, nature and seriousness of observed device malfunctions / deficiencies (DDs).
Time Frame: Day 0 to Day 360 (V01 [Implantation] to V09)
Population: 24 device deficiencies in 14 patients have been documented and were analyzed. The safety and well-being was not affected (or had the potential to affect) in any patient.
Measure: Number; unit: DDs
Units Other Than Participants: DDs
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 24
Number analyzed (DDs) | 24
DDs
  Reader device (external handheld device) | 14
  ARGOS-SC sensor (recalibration of the reader device for compensation, one (1) discontinued use) | 4
  Both reader device and ARGOS-SC sensor | 5
  Other | 1

6. Secondary Outcome: Usability: Implantation Procedure
Description: User acceptance of the ARGOS-SC implantation procedure by means of evaluation of implantation procedure questionnaires (surgeons) on a scale of 1 to 7 how strongly they agree to given statements (1 = totally disagree, 7 = totally agree). Overall Number of Participant Analyzed represents the 7 surgeons who provided feedback via a structured questionnaire. The score 7 represents a greater user acceptance.
Time Frame: Day 1 (V01 [Implantation])
Population: After each implantation procedure, the surgeon performing the implantation procedure was asked to provide feedback on the implantation procedure and the handling of the investigational device. A total of 7 surgeons performed the implantation procedure and provided feedback via a structured questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 7
score on a scale | 6.6 (2.1)

7. Secondary Outcome: Usability: User Acceptance at the Investigational Site
Description: User acceptance of the ARGOS-SC system at the investigational site by means of evaluation of Investigator's questionnaires on a scale of 1 to 7 how strongly they agree to given statements (1 = totally disagree, 7 = totally agree). Overall Number of Participants Analyzed represents the 12 physician investigators who completed the User Acceptance Questionnaire. The score 7 represents a greater user acceptance.
Time Frame: Day 1 to Day 360 (V02 to V09)
Population: The user acceptance questionnaire for physicians was collected from 12 investigators.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 12
score on a scale | 5.5 (3.1)

8. Secondary Outcome: Usability: User Acceptance at Home
Description: User acceptance of the ARGOS-SC system at home by means of evaluation of patient questionnaires on a scale of 1 to 7 how strongly they agree to given statements (1 = totally disagree, 7 = totally agree). The score 7 represents a greater user acceptance.
Time Frame: Day 1 to Day 360 (V02 to V09)
Population: Each patient was asked to provide feedback on the user acceptance of the ARGOS-SC system at home. A total of 19 patients provided feedback via a structured questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGOS-SC Sensor
Number analyzed (Participants) | 19
score on a scale | 5.7 (3.2)

ADVERSE EVENTS:
Time Frame: Evaluation over 12 months follow-up period. Within the timeframe of the ARGOS-SC01 Study: In Germany the term SAE is defined according to §2 Section 5 MPSV.
Description: SAE defined as AE that
  1. Led to death
  2. Led to a serious deterioration in health of a subject that:
     a Resulted in life-threatening illness or injury b Resulted in permanent impairment of a body-structure or function c Required in-patient hospitalization or prolongation of existing hospitalization d Required medical or surgical intervention to prevent permanent impairment to body-structure or a -function
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect
Arm/Group | ARGOS-SC Sensor
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGOS-SC Sensor (N=24)
acute dyspnoe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebral ischemia, left, suspected (Nervous system disorders) | 1 (1)
chronic sleep apnoe (General disorders) | 1 (1)
Hallux Valux Surgery (Surgical and medical procedures) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Stomach ache (Gastrointestinal disorders) | 1 (1)
Syncope (General disorders) | 2 (2)
Syncope, retrograd amnesie and fracture of vertebrae (General disorders) | 1 (1)
intestinak surgery (removal of carcinoma) (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGOS-SC Sensor (N=24)
Conjunctival Wound leak (Eye disorders) | 2 (2)
Endothelium, Erythrocytes (Eye disorders) | 2 (2)
Eye Pain (Eye disorders) | 2 (2)
Hyphema (Eye disorders) | 9 (9) — most common AE was hyphema which was related to medical procedure 7 times in 7 patients, in one patient as probable related to the medical procedure&in another patient as possible related to the medical procedure
Hyposphagma (Eye disorders) | 3 (3)
Reduction of retinal nerve fibre thickness (Eye disorders) | 2 (2)
Secondary Cataract (Eye disorders) | 3 (3)
Thygeson's superficial punctate keratooathy (Eye disorders) | 2 (2)
Touch sensitivity of the eye (Eye disorders) | 3 (3)
Intraocular pressure increased non-study eye (Eye disorders) | 3 (3)
surgical intervention non-study eye (Eye disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03756662/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03756662/SAP_001.pdf